CLINICAL TRIAL: NCT06746714
Title: Testing a New Population Management Model for Hypoglycemia Prevention in High-Risk KPNC Members
Brief Title: Hypoglycemia Prevention in High-Risk Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Lisa K Gilliam, Chief of Endocrinology, South San Francisco Medical Center, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRBNetID: 1980653
Record Dates: First submitted 2024-12-13; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Diabetes
Keywords: hypoglycemia; population management; clinical guideline
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intervention group, receiving protocol-driven outreach by a clinical pharmacist (the "hypoglycemia champion", or HC) to hypoglycemia-prone patients with T2D
  Interventions: Behavioral: Proactive population care (active application of HOAP principles in patients flagged as high risk for hypoglycemia)
- Usual care group (Active Comparator): Usual care, after system-wide dissemination of HOAP
  Interventions: Behavioral: Usual care, after system-side dissemination of HOAP

INTERVENTIONS:
Behavioral: Proactive population care (active application of HOAP principles in patients flagged as high risk for hypoglycemia) — The Hypoglycemia Champion (HC) pharmacist reviewed patient charts before conducting proactive outreach. They did not contact subjects with active psychiatric issues or those admitted to a skilled nursing facility. The patient's care team (PCP and APM) were also contacted for peer consent. The outreach process involved an initial phone call with a secure electronic message or mailed letter (for those without secure KPNC patient portal access) if the initial call was unsuccessful. A second and third phone call attempt was made for non-responders.
  Arms: Intervention group
Behavioral: Usual care, after system-side dissemination of HOAP — Patients had their diabetes treated as usual by their diabetes care provider or primary care physician, after system-wide dissemination of HOAP.
  Arms: Usual care group

SUMMARY:
Severe low blood sugar (hypoglycemia) is a serious problem for people with diabetes. It can lead to dangerous falls, heart problems, memory issues, and even death. However, many healthcare providers don't recognize or manage this problem well. The investigators believe that creating a clear set of guidelines for preventing hypoglycemia, along with having a clinical pharmacist actively help high-risk patients, can make diabetes treatment safer.

In this study, the investigators developed a simple, evidence-based guide called "Hypoglycemia on a Page" (HOAP) to prevent low blood sugars. The investigators then tested it by comparing two groups of patients with type 2 diabetes who are at high risk for hypoglycemia. One group received active support from a clinical pharmacist using the HOAP guidelines, while the other group received standard care.

The main goal of this study is to see if the pharmacist's support leads to safer diabetes treatment. The investigators will also look at other factors, such as whether patients are prescribed glucagon (a medicine for severe low blood sugar), if they use continuous glucose monitoring, and whether they have worse blood sugar control or end up in the hospital for hypoglycemia. This trial aims to improve patient safety, health outcomes, and possibly lower healthcare costs.

DETAILED DESCRIPTION:
The primary research question is whether using a "Hypoglycemia Champion" (HC) to target high risk patients with type 2 diabetes (T2D) is a feasible and effective model of care to reduce hypoglycemia risk in this population.

The goals of this study are to:

1. Develop an evidence-based, expert consensus clinical guideline, "Hypoglycemia on a Page" (HOAP), for hypoglycemia prevention in patients with T2D at high risk of hypoglycemia. Guideline development will include stakeholders across multiple Kaiser Permanente regions.
2. Develop a workflow for use by a "Hypoglycemia Champion" (HC), a clinical pharmacist who will apply the HOAP guideline in the proactive, protocol-driven management of Kaiser Permanente Northern California (KPNC) members identified as having high hypoglycemic risk;
3. Conduct a pragmatic, randomized trial of the proactive HC intervention vs. usual care on diabetes regimen safety among KPNC members at high risk of hypoglycemia. The investigators hypothesize that at 6 months, high-risk members assigned to the HC intervention will be prescribed safer diabetes regimens (defined as discontinuation of sulfonylureas and/or rapid-/short-acting or mixed insulins) compared to usual care.

The study design will include: 1) Engaging expert clinical stakeholders and experienced KP guideline developers to create an evidence-based hypoglycemia prevention algorithm (HOAP) analogous to KPNC's successful "PHASE on a Page" guideline for cardiovascular risk management; 2) Crafting a population-based workflow protocol for proactive outreach by the HC (specifically trained clinical pharmacist) to apply this new guideline to high-risk members; and 3) Performing a pragmatic randomized trial comparing proximal clinical outcomes (diabetes medication changes) available directly from the EHR between the intervention arm (pro-active outreach by the HC) vs. controls (usual care, including availability of the HOAP). The primary analysis will be intent-to-treat and will assess differences in the proportion of patients using safer diabetes regimens (relative to their baseline regimen) between study arms. The investigators will also examine heterogeneity of treatment effects by age, race/ethnicity, and prior severe hypoglycemia events. Deliverables include: 1) Inter-regional dissemination of the HOAP algorithm and the HC workflow protocol, 2) High quality, pragmatic RCT results to inform operational decision-making, and 3) Presentations and manuscripts to further disseminate findings. This study is highly relevant to TPMG and KP because: 1) Hypoglycemia is common, morbid, and costly, 2) Providers are challenged to address the competing demands of prescribing diabetes medications to meet glycemic targets while avoiding iatrogenic hypoglycemia, 3) No regional strategies currently exist to reduce hypoglycemia risk. This work has strategic implications for our organization because a new HEDIS measure proposed for measurement year 2023 will assess emergency department admissions for hypoglycemia in older adults with diabetes. Our proposal will address this gap in organizational clinical care by developing and evaluating a practical, proactive, population management approach to hypoglycemia prevention for members with T2D at high risk of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Active KPNC members with valid MRNs at baseline (06/01/2023),
2. age >=18 years,
3. in the KPNC diabetes registry,
4. likely type 2 diabetes (determined using a validated algorithm
5. high risk for hypoglycemia, determined using the hypoglycemia risk stratification tool developed by the investigator team

Exclusion Criteria:

1. Dementia or impaired cognition,
2. psychosis or schizophrenia diagnosis,
3. end-stage renal disease,
4. "no contact" preferences on file,
5. no primary care physician or home facility,
6. receiving care at skill nursing facilities,
7. deceased,
8. enrolled in concurrent pharmacy deprescribing pilots

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with sulfonylureas, mealtime, or mixed insulin discontinued | 6 months
  We will test for differences in the proportion of patients prescribed safer diabetes regimens (i.e., discontinuation of sulfonylureas, mealtime or mixed insulin)

SECONDARY OUTCOMES:
Number of participants prescribed CGM | 6 months
  We will test for differences in the proportion of patients prescribed CGM
Number of participants prescribed glucagon | 6 months
  We will test for differences in the proportion of patients prescribed glucagon
Number of participants with A1c <8% | 6 months
  We will test for differences in the proportion of patients with good glycemic control (A1c <8%)
Number of participants with ED visit or hospitalization for hypoglycemia | 6 months
  We will test for differences in the proportion of patients who had an ED visit or hospitalization for hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K Gilliam, MD, PhD, Principal Investigator — The Permanente Medical Group
Locations (1):
- Kaiser Permanente Department of Research, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No
The data generated and/or analyzed by the described study are not publicly available due to institutional policies but are available from the corresponding author on reasonable request and with the appropriate IRB approvals.

REFERENCES:
- [Background] Karter AJ, Warton EM, Lipska KJ, Ralston JD, Moffet HH, Jackson GG, Huang ES, Miller DR. Development and Validation of a Tool to Identify Patients With Type 2 Diabetes at High Risk of Hypoglycemia-Related Emergency Department or Hospital Use. JAMA Intern Med. 2017 Oct 1;177(10):1461-1470. doi: 10.1001/jamainternmed.2017.3844. PMID 28828479
- [Background] Schroeder EB, Donahoo WT, Goodrich GK, Raebel MA. Validation of an algorithm for identifying type 1 diabetes in adults based on electronic health record data. Pharmacoepidemiol Drug Saf. 2018 Oct;27(10):1053-1059. doi: 10.1002/pds.4377. Epub 2018 Jan 2. PMID 29292555
- [Background] Klompas M, Eggleston E, McVetta J, Lazarus R, Li L, Platt R. Automated detection and classification of type 1 versus type 2 diabetes using electronic health record data. Diabetes Care. 2013 Apr;36(4):914-21. doi: 10.2337/dc12-0964. Epub 2012 Nov 27. PMID 23193215
- [Background] Parker MM, Moffet HH, Adams A, Karter AJ. An algorithm to identify medication nonpersistence using electronic pharmacy databases. J Am Med Inform Assoc. 2015 Sep;22(5):957-61. doi: 10.1093/jamia/ocv054. Epub 2015 Jun 15. PMID 26078413
- [Background] Karter AJ, Parker MM, Moffet HH, Ahmed AT, Schmittdiel JA, Selby JV. New prescription medication gaps: a comprehensive measure of adherence to new prescriptions. Health Serv Res. 2009 Oct;44(5 Pt 1):1640-61. doi: 10.1111/j.1475-6773.2009.00989.x. Epub 2009 Jun 3. PMID 19500161
- [Background] Moffet HH, Adler N, Schillinger D, Ahmed AT, Laraia B, Selby JV, Neugebauer R, Liu JY, Parker MM, Warton M, Karter AJ. Cohort Profile: The Diabetes Study of Northern California (DISTANCE)--objectives and design of a survey follow-up study of social health disparities in a managed care population. Int J Epidemiol. 2009 Feb;38(1):38-47. doi: 10.1093/ije/dyn040. Epub 2008 Mar 7. No abstract available. PMID 18326513
- [Background] Hui RL, Chang CC, Niu F, Tang YK, Harano D, Deguzman L, Kao DJ, Awsare S, Draves M. Evaluation of a Pharmacist-Managed Antidiabetic Deprescribing Program in an Integrated Health Care System. J Manag Care Spec Pharm. 2019 Aug;25(8):927-934. doi: 10.18553/jmcp.2019.25.8.927. PMID 31347983
- [Background] Kaur U, Machado M, Mistry A. Hypoglycemia: A closer look at a community pharmacist's impact in optimizing diabetes care. J Am Pharm Assoc (2003). 2022 Sep-Oct;62(5):1686-1693.e6. doi: 10.1016/j.japh.2022.04.002. Epub 2022 Apr 12. PMID 35550730
- [Background] Whitfield N, Gregory P, Liu B, Spratt S, Smith BH. Impact of pharmacist outreach on glucagon prescribing. J Am Pharm Assoc (2003). 2022 Jul-Aug;62(4):1384-1388.e1. doi: 10.1016/j.japh.2022.01.017. Epub 2022 Jan 31. PMID 35151583
- [Background] Choe HM, Mitrovich S, Dubay D, Hayward RA, Krein SL, Vijan S. Proactive case management of high-risk patients with type 2 diabetes mellitus by a clinical pharmacist: a randomized controlled trial. Am J Manag Care. 2005 Apr;11(4):253-60. PMID 15839185
- [Background] Lipska KJ, Warton EM, Huang ES, Moffet HH, Inzucchi SE, Krumholz HM, Karter AJ. HbA1c and risk of severe hypoglycemia in type 2 diabetes: the Diabetes and Aging Study. Diabetes Care. 2013 Nov;36(11):3535-42. doi: 10.2337/dc13-0610. Epub 2013 Jul 30. PMID 23900589
- [Background] Kunutsor SK, Balasubramanian VG, Zaccardi F, Gillies CL, Aroda VR, Seidu S, Khunti K. Glycaemic control and macrovascular and microvascular outcomes: A systematic review and meta-analysis of trials investigating intensive glucose-lowering strategies in people with type 2 diabetes. Diabetes Obes Metab. 2024 Jun;26(6):2069-2081. doi: 10.1111/dom.15511. Epub 2024 Feb 26. PMID 38409644
- [Background] Vijayakumar P, Liu S, McCoy RG, Karter AJ, Lipska KJ. Changes in Management of Type 2 Diabetes Before and After Severe Hypoglycemia. Diabetes Care. 2020 Nov;43(11):e188-e189. doi: 10.2337/dc20-0458. Epub 2020 Sep 17. No abstract available. PMID 32943439
- [Background] Zhao Y, Shi Q, Wang Y, Fonseca V, Shi L. Economic burden of hypoglycemia: Utilization of emergency department and outpatient services in the United States (2005-2009). J Med Econ. 2016 Sep;19(9):852-7. doi: 10.1080/13696998.2016.1178126. Epub 2016 May 4. PMID 27074526
- [Background] Lipska KJ, Ross JS, Wang Y, Inzucchi SE, Minges K, Karter AJ, Huang ES, Desai MM, Gill TM, Krumholz HM. National trends in US hospital admissions for hyperglycemia and hypoglycemia among Medicare beneficiaries, 1999 to 2011. JAMA Intern Med. 2014 Jul;174(7):1116-24. doi: 10.1001/jamainternmed.2014.1824. PMID 24838229
- [Background] Shehab N, Lovegrove MC, Geller AI, Rose KO, Weidle NJ, Budnitz DS. US Emergency Department Visits for Outpatient Adverse Drug Events, 2013-2014. JAMA. 2016 Nov 22;316(20):2115-2125. doi: 10.1001/jama.2016.16201. PMID 27893129
- [Background] Karter AJ, Moffet HH, Liu JY, Lipska KJ. Surveillance of Hypoglycemia-Limitations of Emergency Department and Hospital Utilization Data. JAMA Intern Med. 2018 Jul 1;178(7):987-988. doi: 10.1001/jamainternmed.2018.1014. PMID 29710182